CLINICAL TRIAL: NCT06999226
Title: RENEW-AI: Personalizing Scleroderma Management With an AI Health Coach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Nirali Mukesh Shah, Research Fellow, Physical Medicine and Rehabilitation, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HUM00257292
Record Dates: First submitted 2025-05-22; First posted 2025-05-31 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Scleroderma
Keywords: Systemic Sclerosis
MeSH Terms: conditions — Scleroderma, Diffuse; Scleroderma, Systemic

STUDY DESIGN:
Intervention Model Description: Phase 2 will involve a single-arm, pre-post study design where 20 participants of the original RENEW trial will use the NLP-chat feature integrated into the RENEW app over a 4-week period.
Masking Description: The study team members who interact with participants during the enrollment process will be blinded to participant feedback provided during the study to avoid any influence on the participants' experience or outcomes.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RENEW-AI Chat arm (Experimental): Participants (n=20) who participated in the original RENEW trial will get access to a chat functionality within the RENEW app. The chat functionality in the RENEW app is powered by a large language model and tailored using prompt engineering techniques.
  Interventions: Behavioral: RENEW-AI

INTERVENTIONS:
Behavioral: RENEW-AI — AI assisted health coaching using the LLM-driven chat functionality.

SUMMARY:
The purpose of this pilot study is to explore the use of a large language model (LLM) in providing education and behavioral health coaching for individuals with Systemic Sclerosis (SSc). The goal of the LLM is to help user set or modify behavioral goals, provide education, or emotional support as needed by the participant. The primary outcome for this study is to assess the feasibility and acceptability of using an AI-supported health coaching tool over a four-week period.

DETAILED DESCRIPTION:
The study is supported by Dan Barry Trainee Research Program through the Department of Physical Medicine and Rehabilitation at Michigan Medicine.

ELIGIBILITY:
Inclusion Criteria:

* Participants from our previous clinical trial, who received the original RENEW intervention (n=66), will be invited to participate in this study.
* Participants who have a medical diagnosis of systemic sclerosis, any subtype (diffuse, limited, Sine, or overlap)
* Participants who report a mean score 4 or more on the Fatigue Severity Scale, indicative of problematic fatigue; potential mean range 1-9
* Participants who have access to a computer and an internet connection
* Participants who are able to speak and read English.

Exclusion Criteria:

* Individuals who did not participate in the original RENEW trial
* Individuals who lack access to reliable high-speed internet will be excluded to ensure they can fully engage with the AI-supported health coaching and digital components of the study
* Non-English speakers will be excluded because the current version of the AI tool is available only in English
* Individuals planning to initiate any new treatments specifically targeting fatigue, pain, or mood symptoms (such as psychological therapy, structured rehabilitation, or new medications) during the 4-week study period will be excluded, to avoid confounding effects on the study outcomes.
* Individuals with other significant medical or logistical issues that would impede meaningful participation, such as severe concurrent medical conditions, inability to access the RENEW intervention, or cognitive impairments that prevent them from engaging with study procedures, will also be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2025-05-19 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Engagement with the AI chat feature | Up to 4 weeks
  Engagement is measured through app analytics (It will be reported as the proportion of participants who use the chat feature.)
Satisfaction with AI-generated health coaching | 4 weeks
  Satisfaction is self-reported on the mhealth satisfaction survey v 1. It is a 14-item survey with Likert like questions ranging from 1, strongly disagree to 5, strongly agree. Higher scores imply more satisfaction
Acceptability of RENEW | 4 weeks
  Assessed via focus groups

OTHER OUTCOMES:
Change in Fatigue | Baseline, week 4
  Assessed using the Functional Assessment of Chronic Illness Therapy-Fatigue short form (FACIT-F) is a 13 item subscale that allows patient to rate the intensity of their fatigue and its related symptoms on a scale of 0 (not at all) to 4 (very much). The total calculated score varies from 0-52 with a lower score indicating a more severe fatigue level.
Change in Pain interference | Baseline, week 4
  Assessed using the PROMIS Pain Interference short form - 4 item Likert like questions ranging from 1, not at all to 5, very much. Higher scores imply more pain interference
Change in Depressive symptoms | Baseline, week 4
  Assessed using the PROMIS Depression short form - 4 item Likert like questions ranging from 1, never to 5, always Higher scores imply more depression
Change in Resilience | Baseline, week 4
  Assessed using the Connor-Davidson Resilience Scale - 10 item Likert like questions ranging from 0, not true at all to 4, true nearly all the time Higher scores imply more resilience

CONTACTS AND LOCATIONS:
Overall Officials: Nirali Shah, Principal Investigator — University of Michigan; Susan Murphy, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
IPD can be shared upon requests to the PI. Requests will be considered on an individual basis.